CLINICAL TRIAL: NCT05901883
Title: A First-in-Human, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of CEL383 When Administered Intravenously to Healthy Adult Subjects
Brief Title: First-in-human, Single Ascending Dose Study of CEL383 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celsius Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 383-001
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CEL383 Arm (Experimental): Subjects will receive a single intravenous dose of CEL383
  Interventions: Drug: CEL383
- Placebo Arm (Placebo Comparator): Subjects will receive a single intravenous dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CEL383 — Subjects will receive CEL383
  Arms: CEL383 Arm
Drug: Placebo — Subjects will receive placebo
  Arms: Placebo Arm

SUMMARY:
This is a first-in-human, randomized, double-blind, placebo-controlled, single ascending dose study to evaluate the safety, tolerability, and pharmacokinetics of CEL383 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female (of nonchildbearing potential only), 19-64 years of age, inclusive, at screening visit
* Willingness of men of reproductive potential to agree to use a condom with spermicide or abstain from heterosexual intercourse from dosing until at least 90 days after dosing
* Continuous nonsmoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to dosing
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at screening visit
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, and ECGs

Exclusion Criteria:

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study
* History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study
* History or presence of alcohol or drug abuse within the past 2 years prior to dosing
* History or presence of any known primary or secondary immunodeficiency disorder
* History or presence of any signs, symptoms, or diagnosis of infection, including nausea, vomiting, fever, rash, confusion, muscle aches, cough, nasal congestion, or shortness of breath, in the 4 weeks prior to screening or during the screening period.
* History or presence of any known clotting or hemostasis disorder
* Female subject of childbearing potential

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | Through the Day 85 study visit
  Incidence of TEAEs by type, severity, seriousness, and relationship

SECONDARY OUTCOMES:
Cmax | Day 1 through Day 85
  Maximum concentration after single ascending dose
Tmax | Day 1 through Day 85
  Time to reach maximum concentration after single ascending dose
t1/2 | Day 1 through Day 85
  Half-life after single ascending dose
AUC | Day 1 through Day 85
  Area under the curve after single ascending dose
ADA | Day 1 through Day 85
  Incidence of anti-drug antibody after single ascending dose

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Grant, MD, Study Director — Celsius Therapeutics, Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No